CLINICAL TRIAL: NCT03647670
Title: A PHASE 1, RANDOMIZED, 2-WAY CROSSOVER, MULTIPLE DOSE, OPEN LABEL STUDY OF THE EFFECT OF PF-04965842 ON MIDAZOLAM PHARMACOKINETICS IN HEALTHY VOLUNTEERS
Brief Title: A Study to Determine the Effects of PF-04965842 on Midazolam PK in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: B7451022; 2018-001198-26 (EudraCT Number)
Record Dates: First submitted 2018-07-12; First posted 2018-08-27 (Actual); Last update posted 2020-03-23 (Actual); Status verified 2020-03

CONDITIONS: Phase 1
Keywords: PF-04965842
MeSH Terms: interventions — abrocitinib; Midazolam

STUDY DESIGN:
Intervention Model Description: Natural log transformed area under the curve from zero to infinity, area under the plasma concentration-time curve from 0 to the time of last measurement and max plasma concentration of midazolam will be analyzed using a mixed effect model with sequence, period and treatment as fixed effects and subject within sequence as a random effect. Estimates of the adj mean differences (Test-Reference) and corresponding 90% CIs will be obtained from the model. The adjusted mean differences and 90% CIs for the differences will be exponentiated to provide estimates of the ratio of adjusted geometric means (Test/Reference) and 90% confidence intervals for the ratios. Midazolam alone will be the Reference treatment, while the midazolam co-administered with PF-04965842 will be the Test treatment. The lack of an effect of PF-04965842 on midazolam PK will be concluded if the 90% CI for the ratio of adjusted geometric mean for AUCinf falls wholly within acceptance region (80%, 125%).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Sequence 1 (Other): In Sequence 1, Period 1, subjects will be dosed with a single administration of midazolam 2 mg oral solution on Day 1. Midazolam PK will then be assessed over the next 24 hours (hr). Period 1 will be immediately followed by Period 2 with no washout, in which subjects will be dosed with 200 mg PF-04965842 orally once daily (QD) for 7 days. Midazolam 2 mg oral solution will be administered on the morning of Day 2 and Day 7 within 5 minutes after PF-04965842 dosing. Midazolam PK will be assessed for 24 hr following dosing.
  Interventions: Drug: PF-04965842; Drug: Midazolam
- Sequence 2 (Other): In Sequence 2, Period 1, subjects will be dosed with 200 mg PF-04965842 orally QD for 7 days. Midazolam 2 mg oral solution will be administered on the morning of Day 2 and Day 7 within 5 minutes after PF-04965842 dosing. Midazolam PK will be assessed for 24 hr following dosing. Subjects will then undergo a washout period of at least 7 days. In Period 2 subjects will be dosed with a single administration of midazolam 2 mg oral solution on Day 1. Midazolam PK will then be assessed over the next 24 hr.
  Interventions: Drug: PF-04965842; Drug: Midazolam

INTERVENTIONS:
Drug: PF-04965842 — orally bioavailable small molecule that selectively inhibits JAK1 by blocking the adenosine triphosphate (ATP) binding site.
  Other Names: JAK1 Inhibitor
Drug: Midazolam — substrate which undergoes extensive metabolism by CYP3A4 and CYP3A5 and acts as a sensitive probe for evaluating drug interaction with respect to these isoenzymes

SUMMARY:
This is a Phase 1, randomized, 2-way crossover, multiple dose, open label study of the effect of PF-04965842 on midazolam PK in healthy subjects. The study will demonstrate the effect of multiple dose PF-04965842 on the pharmacokinetics of a single, oral dose of midazolam in healthy subjects.

DETAILED DESCRIPTION:
Subjects will be randomized to 1 of 2 treatment sequences as described below. A total of 24 healthy male and/or female subjects will be enrolled in the study so that 12 subjects will be enrolled in each treatment sequence. Each treatment sequence will consist of 2 periods in a single fixed sequence. Subjects will be screened within 28 days of the first dose of study medication. Subjects will report to the clinical research unit (CRU) the day prior to (or Day -1) Day 1 dosing in Period 1 for both treatment sequences. In Sequence 1 subjects will remain in the CRU for a total of 11 days and 10 nights (including Period 1 and Period 2). In Sequence 2, Period 1, subjects will remain in the CRU for 9 days and 8 nights. In Sequence 2, Period 2, subjects will remain in the CRU for 3 days and 2 nights. In Sequence 1, Period 1, subjects will be dosed with a single administration of midazolam 2 mg oral solution on Day 1. Midazolam PK will then be assessed over the next 24 hours (hr). Period 1 will be immediately followed by Period 2 with no washout, in which subjects will be dosed with 200 mg PF-04965842 orally once daily (QD) for 7 days. Midazolam 2 mg oral solution will be administered on the morning of Day 2 and Day 7 within 5 minutes after PF-04965842 dosing. Midazolam PK will be assessed for 24 hr following dosing.In Sequence 2, Period 1, subjects will be dosed with 200 mg PF-04965842 orally QD for 7 days. Midazolam 2 mg oral solution will be administered on the morning of Day 2 and Day 7 within 5 minutes after PF-04965842 dosing. Midazolam PK will be assessed for 24 hr following dosing. Subjects will then undergo a washout period of at least 7 days. In Period 2 subjects will be dosed with a single administration of midazolam 2 mg oral solution on Day 1. Midazolam PK will then be assessed over the next 24 hr.

ELIGIBILITY:
Inclusion Criteria:

* Evidence of a personally signed and dated informed consent document indicating that the subject has been informed of all pertinent aspects of the study
* Willing and able to comply with scheduled visits, treatment plan, laboratory tests and other study procedures
* Healthy female subjects and/or male subjects who, at the time of screening, are between the ages of 18 and 55 years, inclusive
* Female subjects with child-bearing potential must not be intending to become pregnant, currently pregnant, or lactating. Conditions apply: negative pregnancy test, effective method of contraception
* Non-childbearing potential must meet at least 1 of the following criteria: documented hysterectomy and/or bilateral oophorectomy, ovarian failure, achieved postmenopausal status confirmed with FSH
* Body mass index (BMI) of 17.5 to 30.5 kg/m2; and a total body weight >50 kg (110 lbs)

Exclusion Criteria:

* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, GI, CV, hepatic, psych, neurological, or allergic disease (including drug allergies, but excluding seasonal)
* Evidence or history of clinically significant dermatological condition (eg, contact dermatitis or psoriasis) or visible rash present during physical examination
* Subjects, who according to the product label for midazolam, would be at increased risk if dosed with midazolam
* Self-reported history or risk factors for QT prolongation or torsades de pointes, congenital deafness, family history of sudden death, and family history of long QT syndrome
* Any condition possibly affecting drug absorption (eg, gastrectomy)
* A positive urine drug test
* History of regular alcohol consumption exceeding 14 for female or 21 for male drinks/week (1 drink = 5 ounces of wine or 12 ounces of beer or 1.5 ounces of hard liquor) within 6 months of screening
* Treatment with an investigational drug within 30 days (or as determined by the local requirement) or 5 half-lives preceding the first dose of investigational product (whichever is longer)
* Following at least 5 minutes of supine rest, screening supine systolic BP <90 mm Hg or >=140 mm Hg, or screening supine diastolic BP <50 mm Hg or >=90 mm Hg. Any criteria met, BP should be repeated
* Screening supine 12-lead ECG demonstrating: QTcF >450 msec or QRS interval >120 msec. If QTcF exceeds 450 msec, or QRS exceeds 120 msec, the ECG should be repeated
* AST/SGOT or ALT/SGPT >=1.5 × ULN. Total bilirubin level >1× ULN; subjects with a hx of Gilbert's syndrome must have direct bilirubin <= ULN Known relevant history of elevated liver function tests (LFTs)
* History of tuberculosis (TB) (active or latent) or inadequately treated TB infection. Positive QuantiFERON® - TB Gold test
* Any history of chronic infections, any history of recurrent infections, any history of latent infections, or any acute infection within 2 weeks of baseline
* History of disseminated herpes zoster, or disseminated herpes simplex, or recurrent localized dermatomal herpes zoster
* History of sensitivity to heparin or heparin-induced thrombocytopenia
* Pregnant or breastfeeding female; fertile male and WOCBP unwilling to use a highly effective method of contraception through study duration and for at least 28 days after the last dose
* Use of medications and dietary supplements within 7 days or 5 half-lives prior to first dose, acetaminophen/paracetamol <=1 g/day exception. Herbal supplements and hormonal methods of contraception
* Use of tobacco- or nicotine- containing products in excess of the equivalent of 5 cigarettes per day
* Blood donation (excluding plasma donations) of approximately 1 pint (500 mL) or more within 60 days prior to first dose of investigational product
* History of hypersensitivity to midazolam or any other bezodiazapine
* History of HIV, hepatitis B or C; positive testing for HIV, HepBsAg, HepBcAb or HCVAb. As an exception, a positive HepBsAb as a result of subject vaccination is permissible
* Unwilling or unable to comply with the criteria in the Lifestyle Requirements section of this protocol
* Investigator site staff members and their family members, site staff members otherwise supervised by the investigator, or subjects who are Pfizer employees, including their family members
* Other medical or psych condition including active suicidal ideation/ behavior or lab abnormality that the investigator deems inappropriate for this study or may interfere with study results
* Have any malignancies or have a history of malignancies with the exception of adequately treated or excised non-metastatic basal cell or squamous cell cancer of the skin, or cervical carcinoma in situ
* Subjects at significant risk of suicidal or violent behavior

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2018-07-03 (Actual); Primary Completion 2018-10-16 (Actual); Study Completion 2018-10-16 (Actual)

PRIMARY OUTCOMES:
AUCinf of midazolam. | 8 days
  To demonstrate the effect of multiple dose PF-04965842 on the pharmacokinetics of a single, oral dose of midazolam in healthy subjects. The lack of an effect of PF-04965842 on midazolam PK will be concluded if the 90% confidence interval for the ratio of adjusted geometric mean for AUCinf falls wholly within (80%, 125%).

SECONDARY OUTCOMES:
AUClast of midazolam | 8 days
  Adjusted mean differences and 90% confidence intervals for the differences will be exponentiated to provide estimates of the ratio of adjusted geometric means and 90% confidence intervals for the ratios.
Blood Pressure | 8 days
  Number of Subjects with Data of Potential Clinical Concern
Cmax of midazolam. | 8 days
  Adjusted mean differences and 90% confidence intervals for the differences will be exponentiated to provide estimates of the ratio of adjusted geometric means and 90% confidence intervals for the ratios.
Tmax of midazolam. | 8 days
  Adjusted mean differences and 90% confidence intervals for the differences will be exponentiated to provide estimates of the ratio of adjusted geometric means and 90% confidence intervals for the ratios.
t1/2 of midazolam. | 8 days
  Adjusted mean differences and 90% confidence intervals for the differences will be exponentiated to provide estimates of the ratio of adjusted geometric means and 90% confidence intervals for the ratios.
Pulse | 8 days
  Number of Subjects with Data of Potential Clinical Concern
Temperature | 8 days
  Number of subjects with data of potential clinical concern
Adverse Events | 8 days
  Number of Subjects With Treatment-Related Treatment Emergent Adverse Events (TEAEs)
Laboratory tests | 8 days
  Number of Subjects with Laboratory Test Abnormailities

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Clinical Research Unit, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- [Derived] Wang X, Dowty ME, Tripathy S, Le VH, Huh Y, Curto M, Winton JA, O'Gorman MT, Chan G, Malhotra BK. Assessment of the Effects of Abrocitinib on the Pharmacokinetics of Probe Substrates of Cytochrome P450 1A2, 2B6 and 2C19 Enzymes and Hormonal Oral Contraceptives in Healthy Individuals. Eur J Drug Metab Pharmacokinet. 2024 May;49(3):367-381. doi: 10.1007/s13318-024-00893-5. Epub 2024 Mar 30. PMID 38554232
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=B7451022